CLINICAL TRIAL: NCT05867277
Title: The Effect of Music on Nursing Students' Skills, Anxiety, Self-Confidence Perception, Vital Sings
Brief Title: Effect of Music on Nursing Students' Skills, Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Serpil SU, Assistant Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Necmettin E U
Record Dates: First submitted 2023-02-16; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Music
Keywords: Nursing student; intravenous catheter; anxiety; music; self-confidence
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Single-blinded study with parallel groups.
Who Masked: Participant
Masking Description: Participant blinding was performed in this study. Students did not interact with each other while practicing the PIVC placement in different laboratory rooms on the same day. Thus, students were prevented from knowing their group allocation. In addition, when the students received information about the study, they did not know which group they belonged to because they were not informed about the groups. Investigators could not be blinded, as they knew the group allocation of each student group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music (Experimental): Support was received from the Turkish Music Research and Promotion Group (TÜMATA) in choosing the music. To increase attention before and during the PIVC catheter placement skill practice in the intervention group, "Acemaşiran" music was played, which increases the sense of concentration and creativity. To reduce anxiety, "Pentatonic melodies" were played, which gave self-confidence and determination. The music was played from a computer in the vocational skills laboratory using a loudspeaker. During the entire skill practice, the students continued to listen to the music in a light tone.
  Interventions: Other: music
- control (No Intervention): The students in the control group were given standard skills laboratory training without any intervention

INTERVENTIONS:
Other: music — The students in the intervention group listened to music for 15 min before and during the peripheral intravenous catheter placement skill practice.
  Arms: music

SUMMARY:
Objectives: This study aimed to determine the effect of music on nursing students' skills, anxiety, self-confidence perception, and vital signs.

DETAILED DESCRIPTION:
Design: Single-blinded study with parallel groups. Setting: Faculty of Nursing. Participants: Sixty first-year students who took the Nursing Fundamentals course were randomly assigned to the intervention (n = 30) and control (n = 30) groups.

Methods: Data were collected using the Student Information Form, Subjective Self-Confidence Assessment Tool, and State Anxiety Scale from April 6 to 11, 2022. The students in the intervention group listened to music for 15 min before and during the peripheral intravenous catheter placement skill practice, while no intervention was applied in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Taking the Nursing Fundamentals Course for the first time
* Not placing an IV catheter before
* Volunteering to work

Exclusion Criteria:

* Being a healthy vocational high school graduate
* Being a foreign student

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Anxiety evaluated using the State Anxiety Scale | It was applied 10 minutes after the intervention.
  Scores ranging from 20 to 80 points are obtained in the scale.In the total score obtained.
The skill level of the students was evaluated using the "IV Catheter Insertion Skill Checklist" | It was applied 30 minutes after the intervention.
  A minimum of 0 and a maximum of 68 points could be obtained from the checklist.

SECONDARY OUTCOMES:
Students' self-confidence perceptions were determined using a subjective assessment tool. | It was applied 10 minutes after the intervention.
  A score of "0" indicated the lowest self-confidence, and a score of "10" indicated the highest self-confidence.
Blood pressure was evaluated with a sphygmomanometer. | It was measured 10 minutes after the intervention.
  Accepted normal values: Systolic blood pressure: 100-120 mmHg, Diastolic blood pressure: 60-80 mmHg.
Pulse was evaluated with a pulse oximeter device. | It was measured 10 minutes after the intervention.
  Accepted normal values: 60-100 pulse /min
Respiration was evaluated by observation. | It was measured 10 minutes after the intervention.
  Accepted normal values:12-20 respiration /min
Oxygen saturation was evaluated with a pulse oximetry device. | It was measured 10 minutes after the intervention.
  Accepted normal values:SpO2: 95-100%.

CONTACTS AND LOCATIONS:
Overall Officials: Serpil SU, Study Chair — Necmettin Erbakan University
Locations (1):
- Turkey, Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No